CLINICAL TRIAL: NCT02518789
Title: Effects and Mechanism of Pretreatment With Dexmedetomidine to Etomidate Induce Myoclonus During General Anesthesia Induction Period
Brief Title: Effects and Mechanism of Pretreatment With Dexmedetomidine to Etomidate Induce Myoclonus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tangdu-Eto-myo
Record Dates: First submitted 2015-08-03; First posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Myoclonus
Keywords: myoclonus; Etomidate; Dexmedetomidine
MeSH Terms: conditions — Myoclonus | interventions — Dexmedetomidine; Saline Solution; Etomidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low-dose Dexmedetomidine (Experimental): -Pretreatment before anesthesia induction：Intravenous injection dexmedetomidine 0.5 µg/kg，completed within 15 minutes.
  Interventions: Drug: Low-dose Dexmedetomidine; Drug: Etomidate; Drug: midazolam，fentanyl，rocuronium; Drug: propofol，remifentanil，cis atracurium
- High-dose Dexmedetomidine (Experimental): -Pretreatment before anesthesia induction：Intravenous injection dexmedetomidine 1 µg/kg，completed within 15 minutes.
  Interventions: Drug: High-dose dexmedetomidine; Drug: Etomidate; Drug: midazolam，fentanyl，rocuronium; Drug: propofol，remifentanil，cis atracurium
- normal saline Control group (Placebo Comparator): -Pretreatment before anesthesia induction：Intravenous injection normal saline equal quantity，completed within 15 minutes.
  Interventions: Drug: normal saline; Drug: Etomidate; Drug: midazolam，fentanyl，rocuronium; Drug: propofol，remifentanil，cis atracurium

INTERVENTIONS:
Drug: Low-dose Dexmedetomidine — Pretreatment：Intravenous injection dexmedetomidine 0.5 µg/kg ，completed within 15 minutes.
  Other Names: Yisi
  Arms: Low-dose Dexmedetomidine
Drug: High-dose dexmedetomidine — Pretreatment：Intravenous injection dexmedetomidine 1 µg/kg ，completed within 15 minutes.
  Other Names: Yisi
  Arms: High-dose Dexmedetomidine
Drug: normal saline — Pretreatment：Intravenous injection normal saline equal quantity，completed within 15 minutes.
  Other Names: Sodium Chloride Physiological Solution
  Arms: normal saline Control group
Drug: Etomidate — After 90 seconds of Pretreatment，intravenous infusion of etomidate fat emulsion 0.3mg/kg.
  -Does not offer any other drugs within 5 min after completion of etomidate.
  Other Names: Fuerli
Drug: midazolam，fentanyl，rocuronium — Anesthesia induction：Intravenous injection midazolam 0.03 ~ 0.05 mg/kg, fentanyl 5 ~ 8 g/kg, rocuronium 0.6 mg/kg
  Other Names: Liyuexi，Fentanyl Citrate Injection，Aikesong
Drug: propofol，remifentanil，cis atracurium — Anesthesia maintenance：Intravenous infusion of propofol 4 ~ 6 mg/kg/h, remifentanil 0.1 ~ 0.3 μg/kg/min, intermittent intravenous injection of cis atracurium 0.05 ~ 0.1mg/kg
  Other Names: Propofol Injection，Ruifen，Cisatracurium Besylate Injection

SUMMARY:
By observing the difference of plasma homovanillic acid concentrations and brain electrical consciousness monitoring Narcotrend index, study the possible mechanism of influencing Etomidate induced myoclonus with Dexmedetomidine pretreatment during general anesthesia induction period.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent
* American Society of Anesthesiologists (ASA)classification:class I~II;undergoing elective surgery patients
* Aged between 18 and 55, 49-67 kg weight
* Body Mass Index（BMI）： 20-30 kg/m2
* Did not use any analgesic or sedatives drugs within 24 h pre-operation

Exclusion Criteria:

* Recently patients undergoing sedative drugs and antidepressant treatment
* Serious vision, hearing impairment or other reasons can not communicate
* Serious neurological disease, pregnancy, diseases of the cardiovascular system；
* BMI is Less than the standard 80% or higher than the standard 120%

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
myoclonus level | when myoclonus occurs after emulsion injection is completed，assessed up to 5 minutes
  * Level 0 ：no myoclonus happened;
  * Level 1 ：mild, tiny movement, one part of the body such as a finger or shoulder movement;
  * Level 2 ：moderate ,2 pieces of different muscle or slight movement of the muscle groups, such as face or legs;
  * Level 3 ：severely, 2 pieces or more muscle contracture intensity, such as fast outreach of limbs
Plasma homovanillic acid concentration（PHVA） | Measured when myoclonus occurs after emulsion injection is completed，assessed up to 5 minutes; if myoclonus does not appear,measured at 5 minutes after emulsion injection is completed.

SECONDARY OUTCOMES:
Ramsay sedation score | 1 min after entering the operating room; 1 min after dexmedetomidine injection is completed; 1 min after emulsion injection is completed;5 minutes after emulsion injection is completed；
Narcotrend index | 1 min after entering the operating room; 1 min after dexmedetomidine injection is completed; 1 min after emulsion injection is completed;5 minutes after emulsion injection is completed；

CONTACTS AND LOCATIONS:
Overall Officials: LI yumin, PHD, Principal Investigator — Air Force Military Medical University, China

REFERENCES:
- [Background] Schwarzkopf KR, Hueter L, Simon M, Fritz HG. Midazolam pretreatment reduces etomidate-induced myoclonic movements. Anaesth Intensive Care. 2003 Feb;31(1):18-20. doi: 10.1177/0310057X0303100103. PMID 12635389
- [Background] Stockham RJ, Stanley TH, Pace NL, Gillmor S, Groen F, Hilkens P. Fentanyl pretreatment modifies anaesthetic induction with etomidate. Anaesth Intensive Care. 1988 May;16(2):171-6. doi: 10.1177/0310057X8801600207. PMID 3394909
- [Background] Doenicke AW, Roizen MF, Kugler J, Kroll H, Foss J, Ostwald P. Reducing myoclonus after etomidate. Anesthesiology. 1999 Jan;90(1):113-9. doi: 10.1097/00000542-199901000-00017. PMID 9915320
- [Background] Paris A, Philipp M, Tonner PH, Steinfath M, Lohse M, Scholz J, Hein L. Activation of alpha 2B-adrenoceptors mediates the cardiovascular effects of etomidate. Anesthesiology. 2003 Oct;99(4):889-95. doi: 10.1097/00000542-200310000-00022. PMID 14508322
- [Background] Maze M, Virtanen R, Daunt D, Banks SJ, Stover EP, Feldman D. Effects of dexmedetomidine, a novel imidazole sedative-anesthetic agent, on adrenal steroidogenesis: in vivo and in vitro studies. Anesth Analg. 1991 Aug;73(2):204-8. doi: 10.1213/00000539-199108000-00015. PMID 1649559
- [Background] Venn RM, Bryant A, Hall GM, Grounds RM. Effects of dexmedetomidine on adrenocortical function, and the cardiovascular, endocrine and inflammatory responses in post-operative patients needing sedation in the intensive care unit. Br J Anaesth. 2001 May;86(5):650-6. doi: 10.1093/bja/86.5.650. PMID 11575340
- [Background] Mizrak A, Koruk S, Bilgi M, Kocamer B, Erkutlu I, Ganidagli S, Oner U. Pretreatment with dexmedetomidine or thiopental decreases myoclonus after etomidate: a randomized, double-blind controlled trial. J Surg Res. 2010 Mar;159(1):e11-6. doi: 10.1016/j.jss.2009.07.031. Epub 2009 Aug 19. PMID 20018300